CLINICAL TRIAL: NCT07253610
Title: Investigation of the Effects of Bilateral Rectointercostal Fascial Plane Block on Postoperative Acute Pain in Patients Undergoing Laparoscopic Sleeve Gastrectomy
Brief Title: Effect of Bilateral Rectointercostal Fascial Plane Block on Postoperative Pain After Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Istinye Univesitesi HREC
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Pain, Postoperative; Obesity, Morbid; Laparoscopic Sleeve Gastrectomy (LSG); Opioid Use
Keywords: Rectointercostal Fascial Plane Block; Laparoscopic Sleeve Gastrectomy; Morbid Obesity; Opioid Consumption
MeSH Terms: conditions — Pain, Postoperative; Obesity, Morbid | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, double-blind, parallel-group study involving two arms. The RIB group will receive bilateral rectointercostal fascial plane block in addition to standard general anesthesia and intravenous patient-controlled analgesia (PCA), while the control group will receive only general anesthesia and PCA.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind design: Participants and the outcomes assessor were blinded to group allocation. The anesthesiologist performing the block was not blinded due to the nature of the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral Rectointercostal Fascial Plane Block Group (Experimental): Participants in this group will receive bilateral rectointercostal fascial plane (RIB) block under ultrasound guidance prior to induction of general anesthesia. Following surgery, standard intravenous patient-controlled analgesia (PCA) with morphine will be administered.
  Interventions: Other: Bilateral Rectointercostal Fascial Plane Block; Other: Intravenous Patient-Controlled Analgesia (IV PCA) with Morphine
- Control Group (General Anesthesia + PCA) (Active Comparator): Participants in this group will receive only general anesthesia followed by standard intravenous patient-controlled analgesia (PCA) with morphine. No fascial plane block will be performed.
  Interventions: Other: Intravenous Patient-Controlled Analgesia (IV PCA) with Morphine

INTERVENTIONS:
Other: Bilateral Rectointercostal Fascial Plane Block — Under ultrasound guidance, 30 mL of local anesthetic will be injected bilaterally between the rectus abdominis and intercostal muscles at the level of the 6th-7th costal cartilages to achieve rectointercostal fascial plane block prior to general anesthesia.
  Arms: Bilateral Rectointercostal Fascial Plane Block Group
Other: Intravenous Patient-Controlled Analgesia (IV PCA) with Morphine — For all groups, intravenous patient-controlled analgesia (IV PCA) will be initiated in the post-anesthesia care unit (PACU) using a BodyGuard 575 Pain Manager (UK). The total morphine consumption during the first 24 hours postoperatively will be recorded. The PCA regimen will be standardized as follows: no basal infusion, a 1 mg morphine bolus dose, a lock-out interval of 15 minutes, and a maximum dose limit of 10 mg within 4 hours.
  Approximately 45 minutes before the end of surgery, patients will receive 1 g paracetamol, 20 mg tenoxicam, and 3.5 mg morphine intravenously. Postoperatively, paracetamol will be administered every 8 hours and tenoxicam every 12 hours. This postoperative pain management strategy reflects the standard protocol routinely used in our clinic.

SUMMARY:
This randomized controlled study aims to evaluate the effectiveness of the bilateral rectointercostal fascial plane (RIB) block for postoperative pain management in patients undergoing laparoscopic sleeve gastrectomy. The study compares RIB block combined with standard general anesthesia to standard intravenous patient-controlled analgesia alone. The primary outcome is total opioid consumption within the first 24 postoperative hours, while secondary outcomes include pain scores, patient satisfaction, postoperative nausea and vomiting, and block-related complications.

DETAILED DESCRIPTION:
Adequate pain relief in the postoperative period is a crucial determinant of patient comfort, early mobilization, and overall recovery after laparoscopic sleeve gastrectomy. Effective analgesia not only enhances patient satisfaction but also reduces postoperative complications, facilitates respiratory function, and shortens hospital stay. Conversely, inadequate pain control may lead to delayed mobilization, nausea, vomiting, increased opioid requirements, and prolonged recovery.

In recent years, regional anesthesia techniques, particularly abdominal wall and fascial plane blocks, have become an integral part of multimodal analgesia strategies designed to reduce opioid consumption and minimize related adverse effects. The rectointercostal fascial plane (RIB) block, first described by Tulgar et al. in 2023, is a novel regional technique that targets the thoracoabdominal intercostal nerves by injecting local anesthetic between the rectus abdominis and intercostal muscles at the level of the costal cartilage. This block has shown promising results in providing effective postoperative analgesia after upper abdominal laparoscopic surgeries.

The present randomized controlled study was designed to evaluate the effectiveness of the bilateral rectointercostal fascial plane block compared with standard intravenous patient-controlled analgesia in patients undergoing laparoscopic sleeve gastrectomy. The primary outcome is total opioid consumption during the first 24 postoperative hours, and the secondary outcomes include pain scores at rest and during movement, patient satisfaction, incidence of postoperative nausea and vomiting, and block-related complications.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Body mass index (BMI) > 35 kg/m²
* American Society of Anesthesiologists (ASA) physical status II-III
* Scheduled for elective laparoscopic sleeve gastrectomy under general anesthesia
* Provided written informed consent to participate in the study

Exclusion Criteria:

* Chronic opioid use or dependence
* History of chronic pain
* Known allergy or contraindication to local anesthetics or opioids
* Severe cardiac, hepatic, or renal disease
* Severe psychiatric disorder (e.g., psychosis, dementia)
* STOP-BANG score ≥ 5 (high risk for obstructive sleep apnea)
* Block failure or incomplete block after local anesthetic injection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2025-11-01 (Actual); Primary Completion 2025-12-21 (Actual); Study Completion 2025-12-21 (Actual)

PRIMARY OUTCOMES:
Cumulative Opioid Consumption in the First 24 Hours After Surgery | Postoperative day 1 (0-24 hours after surgery)
  The primary outcome is defined as the total cumulative opioid consumption during the first 24 hours after surgery. Opioid use will be recorded as the total amount of morphine administered via intravenous patient-controlled analgesia (PCA). Patients will be instructed to request analgesia through the PCA device whenever their numeric rating scale (NRS) pain score is ≥4. No basal infusion will be used

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University Faculty of Medicine, Medical Park Gaziosmanpasa Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will not be shared because the dataset includes sensitive clinical and perioperative information, and institutional data protection policies do not allow the external release of participant-level data.